CLINICAL TRIAL: NCT05101226
Title: Healthy University Bern Through Yoga - A Worksite Wellness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: Healthy UB through Yoga
Record Dates: First submitted 2021-10-14; First posted 2021-11-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Employee; Worksite; Yoga; Wellness; Intervention; 8 week; Perceived health; Stress; Well-being; Online; In Person

STUDY DESIGN:
Intervention Model Description: The participants will be randomly assigned either to the waiting list control group or the intervention group. The intervention group will be evenly split into the attending the yoga classes in person and attending them online.
Masking Description: The participants know in which group they are, as does the yoga instructor and the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention in person (Experimental): The participants in this group will receive 8 weeks of yoga classes, that they attend in person.
  Interventions: Behavioral: Yoga attended in person
- Intervention online (Experimental): The participants in this group will receive 8 weeks of yoga classes, that they attend online via zoom.
  Interventions: Behavioral: Yoga attended online
- Waiting list control in person (Other): The waiting list control in person group will participate in person in the same yoga classes as the intervention in person group but only after the first group has finished the intervention
  Interventions: Behavioral: Yoga attended in person
- waiting list control online (Other): The waiting list control online group will participate online in the same yoga classes as the intervention online group but only after the first group has finished the intervention
  Interventions: Behavioral: Yoga attended online

INTERVENTIONS:
Behavioral: Yoga attended in person — One or two weekly yoga classes taught and attended in person with a duration of 60 minutes each. The participants can chose if they want to attend one or both classes. The classes will start with a 10 minute Warm Up and a short Meditation, 10 minutes Sun Salutations, 15 minutes standing Asanas, 15 minutes sitting and lying Asanas and 10 minutes Shavasanah and Meditation.
  Arms: Intervention in person; Waiting list control in person
Behavioral: Yoga attended online — One or two weekly yoga classes taught and attended online with a duration of 60 minutes each. The participants can chose if they want to attend one or both classes. The classes will start with a 10 minute Warm Up and a short Meditation, 10 minutes Sun Salutations, 15 minutes standing Asanas, 15 minutes sitting and lying Asanas and 10 minutes Shavasanah and Meditation.
  Arms: Intervention online; waiting list control online

SUMMARY:
This study aims to research the effect of a 8-week long worksite yoga intervention on the perceived health of the University of Bern employees. Furthermore, in light of the current transition to online options, this study will compare the effects of yoga classes attended in person to those attended online.

DETAILED DESCRIPTION:
After giving informed consent, the participants of the study will be randomly assigned to the intervention or waiting list control group. The intervention group will take part in a 8-week long yoga program before the christmas break, while the waiting list control group will receive the same intervention at the beginning of the new year. For both time periods the participants will be randomly assigned to the in person or the online group.

There will be four measurement times when all the participants will be asked to fill out an online questionnaire before and after both implementations of the intervention. The questionnaires include demographic data, perceived health (SF-8), perceived stress (PSS), well-being (BIT), physical activity questionaire (Godin Leisure-Time Exercise Questionnaire) as well as a questionnaire concerning the satisfaction of the intervention after the participants have actively taken part in the yoga intervention.

ELIGIBILITY:
Inclusion Criteria:

* Employee of the University of Bern
* Understanding German
* Ability to participate in 8 yoga classes

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Change in perceived health | 8 weeks
  Perceived health measured with the SF-8 before the intervention and at the end of the intervention. Questionnaire used: Short Form Health Survey, 8 Items, scores range between 0 and 100, higher score means better perceived health (= good)
Change in perceived stress | 8 weeks
  Perceived stress measured with the PSS before the intervention and at the end of the intervention. Questionnaire used: PSS-10, 10 items, scores range between 10 and 50, higher scores mean higher levels of stress (= bad)
Change in well-being | 8 weeks
  Well-being measured with the BIT before the intervention and at the end of the intervention. Questionnaire used: Brief Inventory of Thriving (BIT), 10 items, scores range between 10 and 50, higher scores mean a higher level of well-being (= good)

SECONDARY OUTCOMES:
Stability of change in perceived health | 12 weeks
  Perceived health measured with the SF-8 before the intervention and at the end of the intervention and at the follow up. Questionnaire used: Short Form Health Survey, 8 Items, scores range between 0 and 100, higher score means better perceived health (= good)
Stability of change in perceived stress | 12 weeks
  Perceived stress measured with the PSS before the intervention and at the end of the intervention and at the follow up. Questionnaire used: PSS-10, 10 items, scores range between 10 and 50, higher scores mean higher levels of stress (= bad)
Stability of change in well-being | 12 weeks
  Well-being measured with the Brief Inventory of Thriving (BIT) before the intervention and at the end of the intervention and at the follow up. Questionnaire used: Brief Inventory of Thriving (BIT), 10 items, scores range between 10 and 50, higher scores mean a higher level of well-being (= good)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Nigg, Prof. Dr., Study Director — Institute for Sport and Sportscience, University of Bern
Locations (1):
- Institute of Sport and Sportscience, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No